CLINICAL TRIAL: NCT01155518
Title: Effect of Hypogonadotropic Hypogonadism and Replacement With Clomiphene Citrate and Testosterone on Insulin Sensitivity, Body Composition, Inflammation, Sexual Function and Spermatogenesis in Young Type 2 Diabetic Men
Brief Title: Hypogonadism in Young Men With Type 2 Diabetes
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: lack of funding
Sponsor: State University of New York at Buffalo (Other)
Collaborators: American Diabetes Association (Other)
Responsible Party: Principal Investigator, sandeep dhindsa, Assoc Prof of Medicine, State University of New York at Buffalo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1-10-JF-13
Record Dates: First submitted 2010-06-30; First posted 2010-07-01 (Estimated); Results first posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Hypogonadotropic Hypogonadism; Type 2 Diabetes
Keywords: hypogonadism; diabetes; spermatogenesis; insulin resistance
MeSH Terms: conditions — Hypogonadism; Diabetes Mellitus, Type 2; Diabetes Mellitus; Insulin Resistance | interventions — Testosterone; Clomiphene

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- testosterone (Experimental): intramuscular injections every 2 weeks
  Interventions: Drug: testosterone
- clomiphene (Experimental): oral drug thrice a week
  Interventions: Drug: clomiphene
- placebo for testosterone (Placebo Comparator): placebo for testosterone arm
  Interventions: Drug: placebo
- placebo for clomiphene (Placebo Comparator): oral placebo for clomiphene arm
  Interventions: Drug: placebo
- eugonadal obese (No Intervention): obese men with normal testosterone level
- lean (No Intervention): healthy lean men (control)

INTERVENTIONS:
Drug: testosterone — intramuscular every 2 weeks
  Arms: testosterone
Drug: clomiphene — thrice a week
  Arms: clomiphene
Drug: placebo — intramuscular saline injections every 2 weeks
  Arms: placebo for testosterone
Drug: placebo — oral
  Arms: placebo for clomiphene

SUMMARY:
Low testosterone production, known clinically as hypogonadism, appears to be common complication of type 2 diabetes, affecting one in three diabetic men. Hypogonadism is known to be associated with decreased muscle mass, increased fat mass, increased inflammation and decreased fertility. In this grant, the investigators propose to study the effects of having low testosterone on 1) insulin sensitivity, the ability of the body to handle glucose 2) fat and muscle mass at specific areas of the body 3) expression of mediators of inflammation in the blood 4) semen quality. This study will compare diabetic men (with or without hypogonadism). This study will also evaluate the effect of treatment with clomiphene (a drug that increases testosterone and sperm production) or testosterone in men with diabetes and hypogonadism. The investigators hope that this project will help us understand the state of hypogonadism in young type 2 diabetic men who are in their peak fertility years and give us insights into treatment of this condition. With the rising prevalence of type 2 diabetes in the young, this project may have implications for public health.

DETAILED DESCRIPTION:
This project will study young men with type 2 diabetes. We have shown that half of these men have low testosterone levels. This can lead to 1) Low muscle mass; 2) more fat mass; 3) insulin resistance; 4) low sperm count and 5) increased inflammation (that increases the risk of heart disease). This project will study these consequences in detail and also the possibility of reversing them with treatment. Information from this project will be useful in planning of future studies that will evaluate the effect of treatment of low testosterone on mortality, heart disease and stroke.

ELIGIBILITY:
Inclusion Criteria:

* T2D Males with age 18-40 years

Exclusion Criteria:

1. planning to have children in the next one year
2. Use of androgens, CC, hCG, aromatase inhibitors or over the counter health supplements which contain androgens currently or in the past 6 months;
3. PSA > 4ng/ml, symptoms of severe BPH, prostate nodule or severe enlargement on digital rectal examination or h/o prostatic carcinoma
4. Hemoglobin A1c > 8%
5. Hematocrit > 50%
6. History of obstructive sleep apnea
7. Congestive heart failure
8. Use of thiazolidinediones or exenatide
9. currently suffering from depression, with or without treatment
10. history of severe depression in the past which needed hospitalization
11. currently suffering from foot ulcer, significant periodontal disease or any other chronic infectious condition
12. Coronary event or procedure in the previous 6 months
13. Hepatic disease (transaminase > 3 times normal) or cirrhosis
14. Renal impairment (serum creatinine > 1.5)
15. HIV or Hepatitis C positive status
16. Participation in any other concurrent clinical trial

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2010-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sandeep Dhindsa, MBBS, Principal Investigator — SUNY at Buffalo
Locations (1):
- Millard Fillmore Gates Hospital, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Eugonadal Obese: men with obesity and normal testosterone levels
- Control: lean healthy men with normal testosterone levels
Period: Overall Study
Arm/Group | Testosterone | Clomiphene | Placebo for Testosterone | Placebo for Clomiphene | Eugonadal Obese | Control
Started | 1 | 1 | 0 | 0 | 1 | 2
Completed | 1 | 0 (never started the study) | 0 | 0 | 1 | 2
Not Completed | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: no patients were recruited in 2 arms
Groups:
- Total: Total of all reporting groups
Arm/Group | Testosterone | Clomiphene | Placebo for Testosterone | Placebo for Clomiphene | Eugonadal Obese | Lean | Total
Number analyzed (Participants) | 1 | 1 | 0 | 0 | 1 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 34 (0) | 30 (0) |  |  | 36 (0) | 21 (1) | 30 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 1 | 1 | 0 | 0 | 1 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 |  |  | 1 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Insulin Resistance
Description: To compare the insulin sensitivity as measured by whole body glucose uptake during hyperinsulinemic euglycemic (HE) clamp in young T2D men with and without HH.
Time Frame: 6 months
Population: study terminated
Groups:
- Eugonadal Obese: normal testosterone men
- Normal Lean: control
Arm/Group | Testosterone | Clomiphene | Placebo for Testosterone | Placebo for Clomiphene | Eugonadal Obese | Normal Lean
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Groups:
- Eugonadal Obese: obese men with normal testosterone levels
- Control: healthy lean men with normal testosterone levels
Arm/Group | Testosterone | Clomiphene | Placebo for Testosterone | Placebo for Clomiphene | Eugonadal Obese | Control
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1 | 0/0 | 0/0 | 0/1 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/0 | 0/0 | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/1 | 0/0 | 0/0 | 0/1 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes